CLINICAL TRIAL: NCT02224690
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P; CBD) as Adjunctive Treatment for Seizures Associated With Lennox-Gastaut Syndrome in Children and Adults.
Brief Title: A Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P; CBD) as Adjunctive Treatment for Seizures Associated With Lennox-Gastaut Syndrome in Children and Adults
Acronym: GWPCARE4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1423; 2014-002941-23 (EudraCT Number)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Lennox-Gastaut Syndrome
Keywords: Cannabidiol; CBD; Epidiolex; GWP42003-P
MeSH Terms: conditions — Epilepsy; Lennox Gastaut Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GWP42003-P 20 mg/kg/day Dose (Experimental): Participants received GWP42003-P 20 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P 20 mg/kg/day Dose
- Placebo (Placebo Comparator): Participants received placebo (0 mg/mL CBD), volume matched to the 20 mg/kg/day dose, administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003-P 20 mg/kg/day Dose — GWP42003-P was presented as an oral solution containing 100 mg/milliliter (mL) cannabidiol (CBD) in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Other Names: Cannabidiol; Epidiolex
  Arms: GWP42003-P 20 mg/kg/day Dose
Drug: Placebo — Placebo was presented as an oral solution containing 0 mg/mL CBD in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of GWP42003-P as adjunctive treatment in reducing the number of drop seizures when compared with placebo, in participants with Lennox-Gastaut Syndrome (LGS).

DETAILED DESCRIPTION:
This study was a 1:1 randomized, double-blind, 14-week comparison of 20 milligram [mg] per kilogram [kg] per day [mg/kg/day] of GWP42003-P versus placebo. The treatment period consisted of a 2-week titration period followed by a 12-week maintenance period. The study determined the efficacy, safety and tolerability of GWP42003-P compared with placebo. The dose was recommended by the Data Safety Monitoring Committee (DSMC) after assessment of safety and pharmacokinetic data from Part A of study GWEP1332. The first participants enrolled into this study after the DSMC reviewed the safety data from Part A of study GWEP1332. Following study completion, all participants were invited to continue to receive GWP42003-P in an open label extension (OLE) study (under a separate protocol).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have been male or female aged between 2 and 55 years (inclusive).
* Participant must have had a documented history of Lennox-Gastaut syndrome. This included written documentation of having met electroencephalogram (EEG) diagnostic criteria during the participant's history and evidence of at least 1 type of generalized seizure, including drop seizures (atonic, tonic, tonic-clonic or myoclonic) for at least 6 months.
* Participants had a history of slow (<3.0 Hertz) spike-and-wave pattern in an EEG prior to the enrollment into the baseline period.
* Participants were refractory; that is having documented failures on more than one antiepileptic drug (AED).
* Participant must have been taking 1 or more AEDs at a dose which has been stable for at least 4 weeks prior to screening.
* All medications or interventions for epilepsy (including ketogenic diet and vagus nerve stimulation [VNS]) must have been stable for 4 weeks prior to screening and participant is willing to maintain a stable regimen throughout the study. The ketogenic diet and VNS treatments are not accounted as an AED.

Key Exclusion Criteria:

* Etiology of participant's seizures was a progressive neurologic disease. Participants with tuberous sclerosis were not excluded from study participation, unless there was a progressive tumor.
* Participant had an anoxic episode requiring resuscitation within 6 months of screening.
* Participant had clinically significant unstable medical conditions other than epilepsy.
* Participant had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to screening or randomization, other than epilepsy.
* Participant was currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid based medications (including Sativex®) within the 3 months prior to study entry and was unwilling to abstain for the duration of the study.
* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the Investigational Medicinal Product (IMP), such as sesame oil.
* Participant had been part of a clinical trial involving another IMP in the previous 6 months.
* Participant had significantly impaired hepatic function at screening or randomization (Alanine aminotransferase [ALT] >5 x upper limit of normal [ULN] or total bilirubin [TBL] >2 x ULN) OR the ALT or Aspartate aminotransferase (AST) >3 x ULN and (TBL >2 x ULN or international normalized ratio >1.5). This criterion can only be confirmed once the laboratory results are available; Participants randomized into the study who are later found not to meet this criterion should be withdrawn from the study.
* Any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale in the last month or at screening.
* Participant was taking more than 4 concurrent AEDs.
* Participant was taking corticotropins in the 6 months prior to screening.
* Participant was taking long-term systemic steroids (excluding inhaled medication for asthma treatment) or any other daily medication known to exacerbate epilepsy. An exception was made of prophylactic medication, for example, idiopathic nephrotic syndrome or asthma.
* Participant was taking felbamate, and they had been taking it for less than 1 year prior to screening.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 171 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (17):
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Ames, Iowa
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Rochester, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Winchester, Virginia
- Denekamp, BV Zwolle, Netherlands
- Poland (5):
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Lublin
  - Poznan

REFERENCES:
- [Background] Thiele EA, Marsh ED, French JA, Mazurkiewicz-Beldzinska M, Benbadis SR, Joshi C, Lyons PD, Taylor A, Roberts C, Sommerville K; GWPCARE4 Study Group. Cannabidiol in patients with seizures associated with Lennox-Gastaut syndrome (GWPCARE4): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2018 Mar 17;391(10125):1085-1096. doi: 10.1016/S0140-6736(18)30136-3. Epub 2018 Jan 26. PMID 29395273
- [Derived] Specchio N, Auvin S, Greco T, Lagae L, Nortvedt C, Zuberi SM. Clinically Meaningful Reduction in Drop Seizures in Patients with Lennox-Gastaut Syndrome Treated with Cannabidiol: Post Hoc Analysis of Phase 3 Clinical Trials. CNS Drugs. 2025 Oct;39(10):1025-1036. doi: 10.1007/s40263-025-01201-8. Epub 2025 Aug 7. PMID 40775196
- [Derived] Auvin S, Nortvedt C, Fuller DS, Sahebkar F. Seizure-free days as a novel outcome in patients with Lennox-Gastaut syndrome: Post hoc analysis of patients receiving cannabidiol in two randomized controlled trials. Epilepsia. 2023 Jul;64(7):1812-1820. doi: 10.1111/epi.17618. Epub 2023 Apr 28. PMID 37052803
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230
- [Derived] Privitera M, Bhathal H, Wong M, Cross JH, Wirrell E, Marsh ED, Mazurkiewicz-Beldzinska M, Villanueva V, Checketts D, Knappertz V, VanLandingham K. Time to onset of cannabidiol (CBD) treatment effect in Lennox-Gastaut syndrome: Analysis from two randomized controlled trials. Epilepsia. 2021 May;62(5):1130-1140. doi: 10.1111/epi.16878. Epub 2021 Apr 2. PMID 33797076

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The dose level of 20 milligram (mg) per kilogram (kg) per day (mg/kg/day) was recommended by the GWEP1332 Part A (NCT02091206) Data Safety Monitoring Committee after assessment of safety and pharmacokinetic data. The investigational medicinal product (IMP) was given daily in 2 divided doses (the preferred dosing regimen for antiepileptic drugs).
Groups:
- GWP42003-P 20 mg/kg/Day Dose: Participants received GWP42003-P 20 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the open-label extension (OLE) study, the maintenance period was followed by a 10-day taper (10% per day) period.
- Placebo: Participants received placebo (0 mg/milliliter [mL] cannabidiol [CBD]), volume matched to the 20 mg/kg/day dose, administered orally, half in the morning and half in the evening. To maintain the blinded aspect of the study, participants titrated the placebo dose over 11 days and remained at this dose for the 12-week maintenance period. If the participant did not immediately enter the OLE study, the maintenance period was followed by a 10-day taper (10% per day) period.
Period: Overall Study
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Started | 86 | 85
Safety Analysis Set (Received at least 1 dose of IMP; analyzed as per actual treatment received.) | 86 | 85
Intent to Treat (ITT) Analysis Set (Received at least 1 dose of IMP with at least 1 post-baseline efficacy endpoint measurement.) | 86 | 85
Completed | 72 | 84
Not Completed | 14 | 1
Not completed — Adverse Event | 8 | 1
Not completed — Met Withdrawal Criteria | 4 | 0
Not completed — Use of G-tube | 1 | 0
Not completed — Did not meet eligibility criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.478 (8.685) | 15.284 (9.7945) | 15.381 (9.2264)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 45 | 43 | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline In Drop Seizure Frequency During The Treatment Period
Description: Drop seizures were recorded by the participant or caregiver using an interactive voice response system (IVRS) diary. Drop seizures were defined as the subset of tonic-clonic, tonic or atonic seizures that were reported as drop seizures in the IVRS. Percentage change from baseline was calculated as: (frequency during the treatment period - frequency during baseline/frequency during baseline) * 100. The frequency during each period was based on 28-day averages and calculated as: (number of seizures in the period/number of reported days in the IVRS period) *28. Baseline included all available data prior to Day 1 (28-day average). Negative percentages show an improvement from baseline.
Time Frame: Baseline to End of Treatment (EOT) (Day 99) or Early Termination (ET)
Population: ITT Analysis Set: All randomized participants who received at least 1 dose of IMP and had at least 1 post-baseline efficacy endpoint measurement. Participants were analyzed according to the treatment group to which they were randomized.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 86 | 85
percentage change | -43.90 [-69.62 to 1.93] | -21.80 [-45.72 to 1.74]
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0135, Wilcoxon rank-sum test; Median Difference (Final Values) = -17.21, 95% CI 2-sided [-30.32 to -4.09] — Calculated using the Hodges-Lehmann approach

2. Secondary Outcome: Number Of Participants With a ≥50% Reduction From Baseline in Drop Seizure Frequency During The Treatment Period
Description: Drop seizures were recorded by the participant or caregiver using an IVRS diary. Drop seizures included the subset of tonic-clonic, tonic or atonic seizures that were reported as drop seizures in IVRS. Percentage change from baseline was calculated as per the primary outcome measure.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 86 | 85
Participants | 38 | 20
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel; Calculated using a Cochran-Mantel-Haenszel test stratified by age group (2-5, 6-11, 12-17 and 18-55 years); Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.33 to 4.97]

3. Secondary Outcome: Percentage Change From Baseline In Total Seizure Frequency During The Treatment Period
Description: Total seizures included the sum of all seizures (tonic-clonic, tonic, atonic, clonic, myoclonic, countable partial, other partial and absence seizures) recorded by the participant or caregiver using an IVRS diary. Percentage change from baseline was calculated as per the primary outcome measure. Negative percentages show an improvement from baseline.
Time Frame: Baseline to EOT (Day 99) or ET
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 86 | 85
percentage change | -41.24 [-62.85 to -13.00] | -13.70 [-45.00 to 7.27]
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0005, Wilcoxon rank-sum test; Mean Difference (Final Values) = -21.13, 95% CI 2-sided [-33.26 to -9.37] — Calculated using the Hodges-Lehmann approach

4. Secondary Outcome: Subject/Caregiver Global Impression Of Change Assessment (S/CGIC)
Description: The S/CGIC was used to assess the participant's overall condition on a 7-point scale, using the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse, or very much worse" (1 = very much improved; 7 = very much worse). On Day 1 (prior to starting IMP), the caregiver was asked to write a brief description of the participant's overall condition as a memory aid for the S/CGIC questionnaire at subsequent visits. If both a CGIC and SGIC were completed then the CGIC was used; if only a CGIC was completed then the CGIC was used; if only a SGIC was completed then the SGIC was used. Last visit for endpoints assessed at clinic visits was defined as the last scheduled visit (not including the end of taper or safety follow-up visits) at which participant's last evaluation was performed.
Time Frame: Baseline to Last Visit (Day 99) or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 84 | 85
Participants
  Very Much Improved | 15 | 5
  Much Improved | 14 | 9
  Slightly Improved | 20 | 15
  No Change | 27 | 43
  Slightly Worse | 7 | 9
  Much Worse | 1 | 2
  Very Much Worse | 0 | 2
Statistical Analysis 1: Comparison: GWP42003-P 20 mg/kg/Day Dose vs Placebo; Test type: Superiority; p = 0.0012, Regression, Logistic; Ordinal logistic regression model with treatment group as a fixed factor; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.45 to 4.47] — Odds of participants recording a lower score (improvement) on a continuous scale

ADVERSE EVENTS:
Time Frame: Day 1 through Day 137 (Safety Follow-up)
Description: Safety Analysis Set: All participants randomized to treatment who received at least 1 dose of IMP. Participants were analyzed according to the treatment they received.
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 20/86 | 4/85
Other Adverse Events (participants affected / at risk) | 53/86 | 43/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose (N=86) | Placebo (N=85)
Constipation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Drug level increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Liver function test abnormal (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Seizure cluster (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 1
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose (N=86) | Placebo (N=85)
Diarrhoea (Gastrointestinal disorders) | 16 | 7
Vomiting (Gastrointestinal disorders) | 8 | 14
Constipation (Gastrointestinal disorders) | 5 | 4
Pyrexia (General disorders) | 11 | 7
Fatigue (General disorders) | 5 | 2
Sinusitis (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 6
Decreased appetite (Metabolism and nutrition disorders) | 11 | 2
Somnolence (Nervous system disorders) | 12 | 8
Sedation (Nervous system disorders) | 7 | 1
Convulsion (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days